CLINICAL TRIAL: NCT04808167
Title: Remote Ischemic Conditioning for Protection From Treatment-related Cardiotoxicity in Pediatric and Adolescent Patients Undergoing Hematopoietic Stem Cell Transplantation: a Feasibility Study
Brief Title: Remote Ischemic Conditioning in HSCT
Acronym: RICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-2891
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Hematopoietic Stem Cell Transplantations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Therapeutic Group (Experimental): Therapeutic group receives remote ischemic conditioning.
  Interventions: Device: autoRIC®
- Control Group (No Intervention): Control group does not receive remote ischemic conditioning.

INTERVENTIONS:
Device: autoRIC® — The autoRIC device will be modified by the company from the standard cuff inflation of 200 mmHg to 180 mmHg for the purposes of this study. Three cuff sizes are available from the company: small, medium, and large, correlating to standard adult cuff sizes. The remote ischemic preconditioning cycles will be performed daily by trained research personnel during the preparative regimen through day 0 (see Figure 1), defined as transplantation of stem cells (last preconditioning cycle on day -1). A control group will undergo a similar procedure, however, the cuff will not be inflated.
  Arms: Therapeutic Group

SUMMARY:
This is a feasibility study at a single site, Cincinnati Children's Hospital Medical Center. The hypothesis will be tested using a prospective study design. The purpose of the study is to determine tolerability and safety of remote ischemic conditioning in pediatric and adolescent patients undergoing HSCT, with the goal of a larger trial of efficacy to follow. The secondary purpose is to determine if remote ischemic conditioning will reduce subclinical cardiotoxicity as measured by markers of myocardial injury and stress in patients undergoing HSCT. The study will include multiple blood collections and echocardiograms.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric, adolescent, or young adult patients, 10 years of age or above.
2. Able to tolerate upper arm blood pressure inflation.
3. Participating in the BMT Biorepository (2012-1156).

Exclusion Criteria:

1. Systolic blood pressure >160 mmHg.
2. Previous diagnosis of cardiomyopathy (dilated, hypertrophic, restrictive, myocarditis) or congenital heart disease other than bicuspid aortic valve.
3. Chronic kidney disease as defined as a pre-transplant GFR <80
4. Central line in both upper extremities.
5. Known peripheral vascular disease or vasculitis.
6. Platelet count less than 30,000.
7. Known clotting disorder or hypercoagulability
8. Non-English speaking patients.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Adverse events | 18-24 months from start of enrollment
  Patients undergoing HSCT will tolerate remote ischemic conditioning and there will be no adverse effect on therapeutic efficacy or co-morbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ryan, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided